CLINICAL TRIAL: NCT07327476
Title: Effects Of Oral Ice Chips On Prevention of Chemotherapy Induced Oral Mucositis In Patients With Solid Tumors Treated With 5 Fluorouracil and Methotrexate In Tertiary Care Hospital , Lahore: A Randomize Control Trial
Brief Title: Effect of Oral Ice Chips to Prevent Chemotherapy-Induced Oral Mucositis in Patient With Solid Tumor Treated With 5 Fluorouracil and Methotrexate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Aqsa Noor, MS Nursing Student, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Aqsa Noor
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy Induced Oral Mucositis
Keywords: Cryotherapy; Solid tumor; oral mucositis
MeSH Terms: conditions — Stomatitis | interventions — Cryotherapy; Mouthwashes

STUDY DESIGN:
Intervention Model Description: Control Group (mouth wash only) Intervention Group (Oral ice chips + mouth wash)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Participants in control arm will use standard care as mouth wash only
  Interventions: Behavioral: Standard Oral Care (Mouthwash)
- cryotherapy arm (Experimental): Participant in experimental arm will use ice chips during chemotherapy infusion and standard care as mouth wash also.
  Interventions: Behavioral: Oral Cryotherapy (Ice Chips)

INTERVENTIONS:
Behavioral: Oral Cryotherapy (Ice Chips) — For participants in the experimental group will undergone cryotherapy in the form of oral ice chips. Oral ice chips will be applied in oral cavity of patients by the researcher as followings: 5 minutes before chemotherapy session, participants will begin sucking on ice chips. During chemotherapy, ice chips will be continuously sucked for 5 minutes, followed by a 5-minutes break, after that this process repeated for another 5minutes total time of application of ice is 30 minutes.
  Other Names: Oral cryotherapy
  Arms: cryotherapy arm
Behavioral: Standard Oral Care (Mouthwash) — Participants will receive standard oral care using mouthwash (saline/bicarbonate/chlorhexidine) three times daily after chemotherapy at home.
  Other Names: Standard Oral Care; Mouthwash
  Arms: Control Arm

SUMMARY:
The goal of this randomized controlled clinical trial is to determine whether oral cryotherapy using ice chips can prevent and reduce the incidence and severity of chemotherapy-induced oral mucositis in adult cancer patients receiving 5-fluorouracil and methotrexate chemotherapy regimens.

The main questions it aims to answer are:

Does the application of oral ice chips reduce the severity of oral mucositis compared to routine mouth care alone?

Is there a significant difference in oral mucositis grades between patients receiving oral cryotherapy and those receiving standard mouthwash care?

Researchers will compare the experimental group receiving oral ice chips during chemotherapy plus routine mouthwash care with the control group receiving routine mouthwash care only to evaluate the effectiveness of oral cryotherapy in reducing oral mucositis severity.

Participants will:

Be randomly assigned to either the experimental group (n = 51) or control group (n = 51)

Receive chemotherapy with 5-fluorouracil or methotrexate

Use routine mouthwash (normal saline/sodium bicarbonate/chlorhexidine) at home

Receive oral ice chips during chemotherapy infusion (experimental group only)

Be assessed for oral mucositis severity using the WHO Oral Mucositis Grading Scale before and after the intervention

DETAILED DESCRIPTION:
Chemotherapy-induced oral mucositis is a common and serious side effect among cancer patients receiving chemotherapy. It causes pain, difficulties in eating and speaking, a greater risk of infection, bleeding, distress, and an overall lower quality of life. According to WHO the prevalence of mucositis after chemotherapy is between 20% and 40% of cancer patients receiving standard chemotherapy treatments, with higher rates seen in patients undergoing high- dose chemotherapy where the incidence can reach up to 80%. The goal of oral cryotherapy is to apply local cooling to the tissue of oral mucosa to prevent and minimize the incidence and severity of oral mucositis. This study aim is to assess the level of oral mucositis (OM) among cancer patients who receive chemotherapy before and after the application of oral ice cubes. This study will be conducted by using randomize control design. Patient who are receiving chemotherapy with 5-fluorouracil regimens and methotrexate regimens will be considered as population of this study. Non Probability purposive sampling will be used. Total sample of 102 patients will be taken than randomly assign to experimental group(n=51) and control group(n=51). Ice chips will be applied in the oral cavity of experimental group during chemotherapy and mouth wash (normal saline/sodium bicarbonate/chlorhexidine) use in home. Control group will use only mouth wash(normal saline/sodium bicarbonate/chlorhexidine). The severity of oral mucositis will be assess by using WHO oral mucositis grading scale. All collected information will be analyzed through SPSS version 27. The study will utilize descriptive statistics(mean,standard deviation,frequency and percentage) to analyze the demographic characteristics of the sample. To compare mucositis scores between the experimental and control groups the chi-square test will be used. A significance level of p < 0.05 will be considered statistically significant.The findings of current study will guide the nursing practice to improve and may be significant for cancer patients. The findings can support evidence-based nursing care by incorporating ice chips as a simple, cost-effective, and non- pharmacological intervention in oncology settings. Effective use of ice chips may decrease the need for analgesics and topical treatments, reducing potential side effects and healthcare costs. By minimizing pain and discomfort, the intervention may enhance nutritional intake, oral hygiene, and overall quality of life for chemotherapy patients.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18-60 years.
* Patients treated with 5-Fluorouracil and Methotrexate regimens.
* Patients scheduled for a two-week cycle of chemotherapy.
* Patients able to tolerate ice and able to communicate effectively.

Exclusion Criteria

* Patients with diabetes mellitus, cardiovascular disorders, or any immune- compromised disease.
* Patients with head and neck surgeries, oral or pharyngeal cancer, or any problems in the oral cavity.
* Patients currently enrolled in or who have signed consent for any other clinical studies that could interfere with the desired outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Severity of chemotherapy-induced oral mucositis | Both groups will be assessed for the development and severity of oral mucositis on day 7 and day 14 after chemotherapy using the WHO Oral Mucositis Grading Scale.
  The severity of chemotherapy-induced oral mucositis will be assessed using the World Health Organization (WHO) Oral Mucositis Grading Scale. The scale ranges from Grade 0 to Grade 4, where Grade 0 = no oral mucositis, Grade 1 = soreness/erythema, Grade 2 = ulcers but able to eat solid food, Grade 3 = ulcers with liquid diet only, and Grade 4 = severe ulcers requiring enteral or parenteral nutrition. Higher scores indicate more severe oral mucositis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Article: Effect of Ice Chips on Severity of Chemotherapy Induced Oral Mucositis — https://journals.ekb.eg/article_379333.html
- See also: Article: Oral mucositis & oral health related quality of life in women undergoing chemotherapy for breast cancer in Karachi, Pakistan: A multicenter hospital based cross-sectional study — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0295456
- See also: Article: The Effects of Oral Cryotherapy on Chemotherapy-Induced Oral Mucositis in Patients Undergoing Autologous Transplantation of Blood Stem Cells: A Clinical Trial — https://pmc.ncbi.nlm.nih.gov/articles/PMC4888846/